CLINICAL TRIAL: NCT03864497
Title: Exercise Capacity and Single Photon Emission Computed Tomography in Liver Transplantation Candidates Study
Brief Title: Myocardial Perfusion Imaging in Liver Transplantation Candidates
Acronym: ExSPECT
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, William E Moody, Consultant Cardiologist with a Specialist Interest in Cardiac Imaging, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: CARMS-14536
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Myocardial Perfusion Imaging; Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthotopic liver transplantation candidates: No intervention, imaging test and risk stratification as part of routine clinical care.
  Interventions: Procedure: Myocardial perfusion imaging

INTERVENTIONS:
Procedure: Myocardial perfusion imaging

SUMMARY:
The optimal screening strategy for assessment of coronary artery disease in patients with end-stage liver disease (ESLD) is unclear. Although consensus based guidelines support noninvasive stress testing prior to orthotopic liver transplantation (OLT), no prospective studies are available to inform the clinician on perioperative risk stratification. This observational cohort study was designed to determine the prognostic utility of single photon emission computed tomography (SPECT) imaging in OLT candidates.

DETAILED DESCRIPTION:
Controversy over whether SPECT imaging offers clinical utility in ESLD has been fuelled by conflicting reports on its accuracy to diagnose CAD in this setting. Moreover, there are no studies examining whether SPECT imaging provides any incremental prognostic value beyond functional testing in this high-risk cohort. We sought to determine the relative importance of CV risk factors, functional capacity and SPECT perfusion results as independent predictors of cardiovascular mortality in OLT candidates.

ELIGIBILITY:
Inclusion Criteria:

• Liver transplantation candidates with one or more of the following:

* inability to perform >4 METs by history
* insulin-treated diabetes mellitus
* serum creatinine >152μmol/l
* history of MI, PCI or CABG
* stable angina
* cerebrovascular disease
* peripheral vascular disease

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Contraindication to liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with end-stage liver disease were identified after referral to the Queen Elizabeth Hospital Birmingham for CV risk stratification as part of a pre-transplant screening work-up. Subjects were referred for non-invasive CV risk assessment based on the above criteria.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | 10 years

SECONDARY OUTCOMES:
Major adverse cardiovascular event | 10 years
All-cause mortality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Steeds, MD, Study Director — University Hospital Birmingham NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moody WE, Holloway B, Arumugam P, Gill S, Wahid YS, Boivin CM, Thomson LE, Berman DS, Armstrong MJ, Ferguson J, Steeds RP. Prognostic value of coronary risk factors, exercise capacity and single photon emission computed tomography in liver transplantation candidates: A 5-year follow-up study. J Nucl Cardiol. 2021 Dec;28(6):2876-2891. doi: 10.1007/s12350-020-02126-z. Epub 2020 May 11. PMID 32394403